CLINICAL TRIAL: NCT02470351
Title: Study SEARCH 026Assessment of the HIV CNS Reservoir, Neurological and Neuro-cognitive Effects, and Source of Rebound HIV in CNS in Subjects Participating in Study SEARCH 019
Brief Title: Assessment of the HIV CNS Reservoir, Neurological and Neuro-cognitive Effects, and Source of Rebound HIV in CNS
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nittaya Phanuphak, MD, PhD, Nittaya Phanuphak, MD, PhD, SEARCH Research Foundation
Other Study IDs: SEARCH 026
Record Dates: First submitted 2015-06-02; First posted 2015-06-12 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Acute HIV Infection; HIV CNS Involvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HIV RNA standard quantitation will be completed using the Roche COBAS/Amplicor HIV-1 Viral Load v2.0 assay, with a lower limit of quantitation of 20cps/mL. Single Copy Assay (SCA) HIV RNA quantitation in the setting of ART will be performed using 5-10 ml of CSF. In addition, cell associated HIV-DNA (total, integrated and 2LTR circles in total CD4+ T cells will be assessed at CRC-CHUM.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to describe in depth the CNS, CNS HIV reservoir and CNS viral rebound in consenting SEARCH 019 subjects prior to, during and after the SEARCH 019 study intervention (VHM + ART or ART only), at 1) baseline, 2) end of study intervention and start of ART interruption, 3) viral rebound (if occurring) or mid-way during observed ART interruption, and 4) at the end of ART interruption. Study SEARCH 026 itself does not employ any therapeutic interventions. However, consenting subjects will participate in lumbar puncture, non-contrast MRI + MRS, and neuropsychological testing at at least three and at most four time points. Any of the 15 subjects to be enrolled in SEARCH 019 may consent to study SEARCH 026 participation and hence a maximum of 15 subjects may enroll. As this is a sub-study, data will be shared from study SEARCH 019 and no interventions (venipunctures) will be repeated unnecessarily.

DETAILED DESCRIPTION:
1. Clinical 1.1 Neurological exam: SEARCH employs the AIDS Clinical Trials Group (ACTG)-derived HIV macroneurological examination, a physician rated symptoms assessment of cognitive features typical of HIV-associated neurocognitive disorder (HAND) and peripheral neuropathy.

   1.2 Neuropsychological assessments: SEARCH employs the HIV neurocognitive battery originally developed by Maj et al. designed to minimize cultural bias and tested in Bangkok. All subjects will have the full SEARCH battery as previously published, avoiding evaluations following invasive procedures. All testing is completed by certified nurse-psychometrists. Data are compared to a normative set of 500 HIV-negative, healthy, community dwelling Thais and stratified by age and educational attainment to define standardized z-scores. A psychiatric inventory mirrors that used for RV254 and has broad Thai validity data, and research nurses perform a functional assessment based on the Clinical Dementia Scale.

   1.3 Lumbar puncture: Lumbar punctures are completed per standard clinical procedures using a Sprotte® (pencil-point) needle to minimize complications. Standard assessments of CSF and serum, protein and cell count are completed and approximately 20cc are collected and ultra-centrifuged. Cell pellets of CSF will be cryopreserved for future potential studies, with subject consent. Supernatants are divided into 0.5cc aliquots, and frozen to -80oC on the same day. CSF VDRL/RPR will be assessed at baseline for those with positive serology in SEARCH 019 and in follow-up if a new positive serology is reported in SEARCH 019 or if subject was CSF positive at baseline. Participant hospitalization for any research-related adverse events requiring admission will be arranged, if needed.

   1.4 Neuro-imaging: Imaging studies will be performed at the Chulalongkorn University Hospital which is 100 meters from the TRCARC in Bangkok. These studies will take up to one hour maximum MRI scanner time for each subject and may include brain MRI, MRS, DTI and resting state functional MRI (fMRI). MRI and MRS are non-invasive methods to detect brain pathology (MRI) and to determine the in-vivo concentration of brain metabolites (MRS). DTI is a sensitive non-invasive magnetic resonance technique to analyze the three-dimensional diffusion of water within brain tissue. The diffusion of water within the brain is highly dependent on the underlying micro-architecture of the surrounding tissue, which is affected by both normal physiological processes (such as aging) as well as local neuropathological disease processes, such as those seen with HIV infection. Resting state functional MRI (fMRI) reveals patterns of activation of brain networks and is a sensitive measure of brain function prior to structural and anatomical changes detected by other methods. Gadolinium will not be used for research purposes.
2. Laboratory (all pertaining to CSF)

2.1 Measurement of soluble markers: Commercial ELISA kits (Human Quantikine ELISA kits; R&D Systems, Inc.) and Millipore Luminex assays will be used following manufacturer's instructions at the Yale Immune Monitoring Core Laboratory. Soluble biomarkers associated with immune activation and neurocognitive impairment will be measured, including CSF neopterin, MCP-1, sCD14, IL-6, sCD163, and IP-10.

2.2 CSF virology Assays: HIV RNA standard quantitation will be completed using the Roche COBAS/Amplicor HIV-1 Viral Load v2.0 assay, with a lower limit of quantitation of 20cps/mL. Single Copy Assay (SCA) HIV RNA quantitation in the setting of ART will be performed using 5-10 ml of CSF. In addition, cell associated HIV-DNA (total, integrated and 2LTR circles in total CD4+ T cells will be assessed at CRC-CHUM.

2.3 TCR repertoire and avidity of HIV-specific CD8+ T cells in CSF: These may be measured in a subset of samples at VGTI Florida. For the repertoire assay, CSF cell pellets will be polyclonally expanded, and the TCR repertoire will be determined followed by TCR sequencing as previously described. For TCR avidity, T cell clones corresponding to the dominant clonotypes will be generated in vitro to measure their functional sensitivity. The HIV-specific CD8+ T cells clones generated by expansion in the presence of PHA, IL-2 and irradiated feeders will be sequenced for their TCR and will be tested for their TCR functional sensitivity.

2.4 Management of Subjects Resuming ART: If the decision is made to reinitiate ART as per SEARCH 019 ART resumption criteria, then the study visit before ART resumption will be considered this study's final visit and all procedures scheduled for end of study will be conducted at that visit.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers recruited to participate in this study must satisfy all of the inclusion and exclusion criteria for study SEARCH 019.

Exclusion Criteria:

* Subject is pregnant or breast-feeding.
* Any contraindication to lumbar puncture, such as history of bleeding diathesis or known cerebral mass lesion
* Any contraindication to MRI or MRS such as an implanted pacemaker, some older intracranial aneurysm clips, cochlear implants, certain prosthetic devices, implanted drug infusion pumps, neurostimulators, bone-growth stimulators, certain intrauterine contraceptive devices, or any other type of iron-based metal implants. MRI is also contraindicated in the presence of some internal metallic objects such as bullets or shrapnel, as well as most surgical clips, pins, plates, screws, metal sutures, or wire mesh.
* Subject has been diagnosed with a serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with his or her ability to adhere to study requirements or to give informed consent.
* Subject has active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with his or her ability to adhere to study requirements or to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any of the 15 subjects to be enrolled in SEARCH 019 may consent to study SEARCH 026 participation and hence a maximum of 15 subjects may enroll.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
CSF vs. plasma HIV viral load in VHM+ART and ART alone | 34 weeks
  Difference between CSF vs. plasma HIV viral load in VHM+ART and ART alone groups at study baseline (prior to VHM initiation), at time just before ATI, midway through ATI period (if not preceded by viral rebound) and at viral rebound or end of ATI observation period. Unit of measure: copies/mL.
Establishment of HIV in the CNS and the source of resurgent CSF HIV RNA between plasma and CSF variants prior to ART and after VHM intervention. | 34 weeks

SECONDARY OUTCOMES:
Change in levels over time of CSF neopterin (nmol/L), sCD14 (ng/mL), CSF MCP-1 (pg/dL), IP-10 (nmol/L), sCD163 (ng/mL), IL-6 (pg/mL), and HIV RNA (copies/mL) value by single copy assay | 34 weeks
Change over time in appearance of structural and T2 MRI scans including evidence of neuroinflammatory lesions | 34 weeks
Change over time in concentrations of creatine (Cr) of choline (Cho), myoinositol (mI), and n-acetylaspartate (NAA) in the basal ganglia, occipital grey matter, and frontal white matter. Unit of measure of all metabolites is mM. | 34 weeks
Measurement ratios with respect to creatinine (Cr) of choline (Cho), myoinositol (mI), and n-acetylasparate (NAA) in the basal ganglia, occipital grey matter, and frontal white matter. Unit of measure for all metabolites is mM. | 34 weeks
Change over time in measures of fractional anisotropy on diffusion tensor imaging (DTI) in whole brain and voxel-based analysis | 34 weeks
Measurement of mean diffusivity on diffusion tensor imaging (DTI) in whole brain and voxel based analysis. | 34 weeks
Change over time in patterns of functional MRI activity between major brain networks | 34 weeks
Change over time in performance on neuropsychological test battery | 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya - Phanuphak, MD, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- SEARCH Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided